CLINICAL TRIAL: NCT06455865
Title: Efficacy of TPACK Framework-Based Instruction in a Network Information Resources Retrieval and Usage Course: A Quasi-Experiment Among Master's Degree Nursing Students
Brief Title: Efficacy of TPACK-Based Instruction in an Information Resources Course for Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Tao (Other)
Responsible Party: Sponsor-Investigator, Xu Tao, Principal Investigator, Hangzhou Normal University
Organization: Hangzhou Normal University (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 2024XG0014
Record Dates: First submitted 2024-06-03; First posted 2024-06-12 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Smart Classroom; Nursing Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The intervention group received instruction based on the TPACK (Technological Pedagogical Content Knowledge) framework, incorporating a blended learning approach that combined online and offline methods. The curriculum included the same fundamental theories and skills as the control group but integrated digital tools and resources. Online components consisted of interactive MOOC videos, online assignments, peer assessments, and real-time virtual discussions via platforms like DingTalk. Offline components included traditional face-to-face classroom sessions, hands-on practice, group discussions, and collaborative projects. The blended approach aimed to enhance students' engagement and understanding by leveraging technology to facilitate a more interactive and flexible learning experience.
  Interventions: Other: TPACK-Based Blended Learning Instruction
- control group (No Intervention): The control group employed traditional in-person teaching methods, including face-to-face classroom instruction, reading from printed textbooks, and completing homework assignments. The curriculum covered the fundamental theories and skills related to information resource retrieval and usage but did not specifically utilize the TPACK framework. Students primarily received lectures and guidance from the instructor during class and completed assignments and learning tasks independently after class.

INTERVENTIONS:
Other: TPACK-Based Blended Learning Instruction — The control group employed traditional in-person teaching methods, including face-to-face classroom instruction, reading from printed textbooks, and completing homework assignments. The curriculum covered the fundamental theories and skills related to information resource retrieval and usage but did not specifically utilize the TPACK framework. Students primarily received lectures and guidance from the instructor during class and completed assignments and learning tasks independently after class.
  Other Names: experimental group
  Arms: experimental group

SUMMARY:
Study Purpose The purpose of this study is to evaluate the effectiveness of a blended teaching approach based on the TPACK framework in improving the skills of master's degree nursing students in retrieving and using network information resources. The TPACK framework integrates Technology, Pedagogy, and Content Knowledge to enhance teaching and learning experiences.

Study Content and Implementation Plan

This study involves a combination of online and offline teaching methods to help nursing students better understand and utilize various information resources. The main components of the study include:

1. Knowledge Mastery Survey: Students will be assessed on their understanding of the course content using a specially designed survey.
2. Resource Effectiveness Evaluation: The study will measure how helpful students find the different resources used in the course, such as videos, PPTs, and assignments.
3. Skill Improvement Assessment: The study will evaluate the extent to which the course helps improve students' abilities in areas like literature search, document management, and academic writing.
4. Student Satisfaction Survey: Students will provide feedback on their satisfaction with the course through a comprehensive survey.

By implementing these measures, the study aims to minimize any negative effects on students and maximize their learning outcomes in a safe and supportive environment.

DETAILED DESCRIPTION:
This study evaluates the effectiveness of a TPACK (Technological Pedagogical Content Knowledge) framework-based instructional approach in a course on Network Information Resources Retrieval and Usage among master's degree nursing students. The research employs a quasi-experimental design to compare the outcomes of an intervention group, which receives TPACK-based blended learning, with a control group that experiences traditional face-to-face instruction.

This study aims to provide evidence on the efficacy of the TPACK-based blended learning approach in enhancing educational outcomes in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Master's degree students enrolled in the nursing program at the participating university.
* Students who have completed the prerequisite courses relevant to the Network Information Resources Retrieval and Usage course.
* Students who have provided written informed consent to participate in the study.
* Students with regular access to the internet and necessary technological devices for participating in online components of the course.

Exclusion Criteria:

* Students who have previously completed a similar course or have extensive prior experience with network information resources retrieval and usage.
* Students who are unable to commit to the course schedule and requirements due to personal or professional reasons.
* Students with known learning disabilities or conditions that might interfere with their ability to complete the course assessments, unless they receive appropriate accommodations.
* Students who withdraw consent at any point during the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-11-19 (Estimated); Study Completion 2024-12-19 (Estimated)

PRIMARY OUTCOMES:
Mastery of knowledge | 3 monthes
  The Knowledge Mastery Scale was used to evaluate students' knowledge mastery. Through a process of revision informed by the course objectives and content, a final version consisting of 12 items was developed. Participants rated their level of mastery based on their course experiences, with higher scores indicating greater mastery. Example item: "Please evaluate your level of mastery of the course content based on your personal experiences. Choose the option that best reflects your understanding on a scale of 1 to 5."

SECONDARY OUTCOMES:
Effectiveness of resources | 3 monthes
  To find out how much the students perceived the resources used in the course to be helpful in understanding and mastering the course content. The questionnaire was based on a 7-point Likert scale, with scores from 1 to 7 indicating "very unhelpful", "unhelpful", "rather unhelpful", "average", "fairly helpful", "helpful", and "very helpful", with higher scores indicating that the higher the score, the more helpful the resource is perceived by the students.

OTHER OUTCOMES:
Learning satisfaction | 3 monthes
  The Learning Satisfaction Scale was adopted as a student self-assessment scale with 24 entries, containing course satisfaction, teaching satisfaction, platform satisfaction, expected service satisfaction, perceived service satisfaction and overall satisfaction. We adjusted the dimensional entries to match the course content, resulting in a 17-entry satisfaction scale. Participants rated their satisfaction level on a 5-point Likert scale, ranging from "very dissatisfied" to "very satisfied."

CONTACTS AND LOCATIONS:
Overall Officials: Tao Xu, Study Chair — Hangzhou Normal University
Locations (1):
- Hangzhou Normal University, Hangzhou, Zhejiang, China